CLINICAL TRIAL: NCT01690611
Title: Sensory Treadmill to Improve of Balance During Walking
Brief Title: Visual Feedback to Improve Balance During Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, John Jeka, Professor, Temple University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 366151-1
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Other Fall; Patient Falls
Keywords: Balance Training; Walking; Falls
MeSH Terms: interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking & Visual Feedback (Experimental): Individuals in this arm will walk on a treadmill while viewing real time visual feedback regarding their body motions and use the visual feedback to correct their body motions.
  Interventions: Procedure: Treadmill Walking; Other: Visual Feedback
- Walking & No Visual Feedback (Active Comparator): Individuals in this arm will walk on a treadmill without viewing real time visual feedback regarding their body motion.
  Interventions: Procedure: Treadmill Walking

INTERVENTIONS:
Procedure: Treadmill Walking — Individuals will walk at a "comfortable speed" on a treadmill without holding on to the hand rails.
Other: Visual Feedback — Real time feedback regarding body motion while walking.
  Arms: Walking & Visual Feedback

SUMMARY:
The goal of this research is to determine if real time visual feedback of body movements improves balance control more than walking on a treadmill alone. Individuals participating in this research study will be tested using a battery of clinical strength and balance assessments twice before a 4 week training period and once after the training period. The 4 week training period will consist of 12 sessions walking on a treadmill. The experimental group will see real time visual feedback regarding their body movements, and the control group will not receive this visual feedback. Following the 4 week training each participant will again be tested using the battery of clinical strength and balance assessments.

ELIGIBILITY:
Inclusion Criteria:

* Fall Prone Older Adults (history of falls or loss of balance)
* ability to walk on the treadmill hands-free without assistance
* Mini-Mental Status Exam > 23

Exclusion Criteria:

* Current enrollment in physical rehabilitation of any kind
* Medically unstable

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in BESTest Score, A clinical assessment of balance | Tested at 0, 4, and 8 weeks
  Balance Evaluation System Test (BESTest)
Change from Baseline in Berg Balance Test Score | Test will be given at 0, 4, and 8 weeks
Change from Baseline in Activity Specific Balance Confidence Score | Tested at 0, 4, and 8 weeks
  Questionnaire rating balance confidence
Change from Baseline in 6 Minute Walk Test | Tested at 0, 4, and 8 weeks
Change from Baseline in Comfortable Walking Speed | Measured daily, up to 12 days
  This value is determined for each training session

SECONDARY OUTCOMES:
Change from Baseline in Muscle Strength | Tested at 0, 4, and 8 weeks
  Strength of major muscles in the legs and trunk will be measured
Change from Baseline in Overground Walking Speed | Tested at 0, 4, and 8 weeks
Change from Baseline in Center of Mass variability | Tested daily, up to 12 days
  This measure is derived from recorded body position during each training repetition for each of up to 12 days of training.
Change from Baseline in Power spectral density | Tested daily, up to 12 days
  This measure is derived from recorded body position during each training repetition for each of up to 12 days of training.
Change from Baseline in Single/Dual Tasking ability | Tested at 0, 4, and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Jeka, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Collington Episcopal Life Care Community, Mitchellville, Maryland
  - Pearson Hall, Temple University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Anson E, Thompson E, Karpen SC, Odle BL, Seier E, Jeka J, Panus PC. Visual biofeedback training reduces quantitative drugs index scores associated with fall risk. BMC Res Notes. 2018 Oct 22;11(1):750. doi: 10.1186/s13104-018-3859-7. PMID 30348198